CLINICAL TRIAL: NCT05392491
Title: The Brazilian Coronary Disease Cohort
Brief Title: Brazilian Coronary ARtery Disease
Acronym: BARD
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BARD Study
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Outcomes; Cohort
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control group (without coronary lesions): Cohort control group. No interventions.
  Interventions: Other: No intervention
- Coronary Lesion < 30%: Participants with coronary lesion under 30%. No interventions.
  Interventions: Other: No intervention
- Coronary Lesion > 30% and < 50%: Participants with coronary lesions greater than 30% and under 50%. No interventions.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention. It is an observational study

SUMMARY:
Although coronary artery disease may have a stable chronic clinical course, it is known that this reality does not apply to atherosclerotic plaques, they can grow, complicate, stabilize and again start new cycles of growth/destabilization/stabilization or quiescence in the presence or absence of symptoms. While in obstructive coronary lesions there are well-founded guidelines based on multiple clinical studies, in relation to investigation and treatment; on the other hand, in non-obstructive lesions, there are no such guidelines. There are gaps in the knowledge about the prognostic implications of minor injuries and the occurrence of events. This study seeks precisely to fill these knowledge gaps. Of particular relevance are the large number of patients (approximately 10,000 patients) and the long clinical follow-up, that is, in eight years.

DETAILED DESCRIPTION:
Introduction:

For decades, patients with obstructive coronary disease, specifically with lesions above 70%, have been the subject of numerous randomized studies and meta-analyses concerning the influence of drug treatments, revascularization (surgical or percutaneous), and lifestyle on their prognosis. In this scenario, the investigators already have a reasonable knowledge of the behaviors most appropriate for both avoiding events and alleviating symptoms. However, one particular subgroup consists of patients whose lesions are non-obstructive. In most cases, these are considered lesions of ≤70%. Many individuals presented obstructive lesions that were deemed appropriate for angioplasty within this classification. For example, in the study Defer of 325 patients with indications of ischemia, 44.3% presented FFR (fractional flow reserve) ≤0.75, which suggested significant obstruction, and were submitted to ATC. Thus, the investigators consider the threshold ≤70% inappropriate since it includes many patients with ischemia when assessed by FFR. Therefore, this study has decided to investigate patients with lesions of ≤50% on the supposition that they do not have obstructive lesions. In addition, although coronary disease may follow a stable clinical course, this is not the case with atherosclerotic plaques. These can grow, become complex, stabilize and reinitiate new cycles of growth/destabilization/stabilization or inactivity, in either the presence or absence of evident symptoms. Though aware of this dynamic, studies were performed to "photograph" at a given time subclinical atherosclerotic load and correlate it to the incidence of the events. The indicators most used for evaluating atherosclerotic load have been the presence of extra-cardiac atherosclerosis (carotid ultrasound) and calcification of the coronary arteries. Furthermore, the calcium score has been used for the same purpose in the Brazilian population: but only as a prognostic indicator among carriers of family hypercholesterolemia. However, there are considerable doubts concerning therapeutic interventions in asymptomatic patients with no critical stenosis. Given this gap, chiefly among the Brazilian population, and being an institution with one of the highest volumes of medical care and screening for coronary disease globally, the investigators have all the necessary conditions to put this important public health problem into perspective.

Objectives:

To evaluate clinical evolution, in eight years, of patients with no coronary lesions or lesions <50%, invasive coronary angiography (ICA) exams or coronary angiotomography is performed for the diagnosis of coronary disease.

Population:

Patients were referred to Instituto do Coração (InCor HCFMUSP) for ICA or angiotomography for diagnosis of coronary heart disease from January 1, 2011, to December 31, 2017. Exclusion criteria: age under 18 years or over 80 years at the time of examination, previous history of an acute coronary syndrome (infarction and unstable angina), revascularization interventions (surgical or percutaneous), valvular heart disease, cardiomyopathies, or diseases with a poor prognosis (expected survival of fewer than eight years). The cohort will be composed of 3 groups: the control group (without coronary lesions), lesion group <30%, and lesion group >30% to <50%. Study type: an observational, retrospective, with data from the database of InCor, (Heart Institute - InCor, University of São Paulo). Outcomes: primary composite (general death, acute myocardial infarction, cerebrovascular accident, need for revascularization); secondary outcomes: the isolated components of the primary outcome at eight years.

Data to be collected:

Age (on the date of examination), gender, presence of risk factors - arterial hypertension (BP >130/85; or use of antihypertensive medication), diabetes mellitus (fasting glucose ≥126 mg/dL, casual >140 mg/dL or GTT >200 mg/dL, or use of oral or injectable hypoglycemic agents), dyslipidemia (LDL >130 mg/dL, triglycerides >150 mg), lipid levels (total cholesterol, HDL-C, LDL-C, and triglycerides); tobacco user (never, ex-tobacco user, active), obesity, exercise, family history, creatinine, chronic kidney disease (glomerular filtration <60 mL/1.73m²/min).

Medications in use: ACE inhibitors/ARB; statins; AAS; Beta-blockers and calcium channel antagonists, and diuretics.

Clinical status: angina and/or dyspnea. Left ventricular systolic function: normal left ventricular ejection fraction (LVEF) (50%), mild decrease (≥45% to <50%); moderate (>35% to 45%) and severe (<35%).

Cardiovascular history: cerebrovascular accident or peripheral arterial disease.

Atherosclerotic load: a) Higher percentage of obstruction of the lumen by comparing the diameter in the lesion region with its proximal neighborhood: absent (0%), very mild (1-30%), and mild (30-49%), for eligibility of each group studied; b) Total lesion score: zero for absence, 1 for minor injuries(<30%), and 2 for minor injuries(30-50%). Multiplied by their frequency and totaled at the end; c) The atherosclerotic load will be weighted using the Syntax scores for its location, though the lesions are less than 50%. Left coronary trunk = 5; proximal AD = 3.5; medial AD = 1.5; distal AD = 1; diagonal = 1; proximal circumflex = 1.5; distal = 1; marginal = 1; proximal or distal right coronary artery = 1 and posterior descending artery = 1; coronary calcium score (CAC).

Population:

Patients underwent invasive coronary angiography (ICA) or coronary computed tomography angiography at InCor from January 2011 to December 2014. To allow 5-year follow-up (FU) of all cases. The investigators estimate the inclusion of approximately 5,000 patients, with a minimum of 1,500 in the control group.

Deadlines for execution and analysis:

The investigators anticipate including an average of 40 patients per day and completion at the end of 2 years. The rate of scheduled events should not exceed 0.5% to 1% per year, so the investigators plan interim analyses at two years FU when the investigators would have at least 600 events for analysis.

Clinical, laboratory, and image data:

Electronic Patient Care System SI3 of InCor will be used to screen and follow the patients. Patients who have not been followed regularly at ambulatory clinics of InCor will be contacted by phone or e-mail to ascertain their evolution. In cases of death, family members or attending physicians will be contacted. Death certificates will be analyzed to adjudicate death´s causes. Eventually, the Foundation for the State System of Data Analysis (SEADE) database from Estado de São Paulo will be used.

ELIGIBILITY:
Inclusion Criteria:

• Patients referred to Instituto do Coração (InCor HC, FM-USP) for invasive coronary angiography or angiotomography.

Exclusion Criteria:

* Age under 18 years or over 80 years at the time of examination;
* Previous history of acute coronary syndrome (infarction and unstable angina);
* Revascularization interventions (surgical or percutaneous);
* Valvular heart disease;
* Cardiomyopathies;
* Diseases with a poor prognosis (expected survival of less than 8 years).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to Instituto do Coração (InCor HC, FM-USP) for invasive coronary angiography or angiotomography, for diagnosis of coronary heart disease from January 1, 2011 to December 31, 2017.
Sampling Method: Non-Probability Sample
Enrollment: 4004 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with Composite Outcome | 8 years
  Participants presenting the following outcomes: death of any cause, acute myocardial infarction, stroke, and need for revascularization.

SECONDARY OUTCOMES:
Number of participants with acute myocardial infarction | 8 years
  According to classical definition: clinical, electrocardiography and enzymes
Number of participants with stroke | 8 years
  Loss of consciousness and hemiplegia
Number of participants needing revascularization | 8 years
  Coronaries bypass surgery or angioplasty

CONTACTS AND LOCATIONS:
Overall Officials: Protasio Luz, PhD, Principal Investigator — Instituto do Coração InCor, Hospital das Clínicas HCFMUSP, Faculdade de Medicina, Universidade de São Paulo
Locations (1):
- Instituto do Coração InCor, Hospital das Clínicas HCFMUSP, Faculdade de Medicina, Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makarovic Z, Makarovic S, Bilic-Curcic I, Mihaljevic I, Mlinarevic D. NONOBSTRUCTIVE CORONARY ARTERY DISEASE - CLINICAL RELEVANCE, DIAGNOSIS, MANAGEMENT AND PROPOSAL OF NEW PATHOPHYSIOLOGICAL CLASSIFICATION. Acta Clin Croat. 2018 Sep;57(3):528-541. doi: 10.20471/acc.2018.57.03.17. PMID 31168187
- [Background] Maddox TM, Stanislawski MA, Grunwald GK, Bradley SM, Ho PM, Tsai TT, Patel MR, Sandhu A, Valle J, Magid DJ, Leon B, Bhatt DL, Fihn SD, Rumsfeld JS. Nonobstructive coronary artery disease and risk of myocardial infarction. JAMA. 2014 Nov 5;312(17):1754-63. doi: 10.1001/jama.2014.14681. PMID 25369489
- [Background] Bech GJ, De Bruyne B, Pijls NH, de Muinck ED, Hoorntje JC, Escaned J, Stella PR, Boersma E, Bartunek J, Koolen JJ, Wijns W. Fractional flow reserve to determine the appropriateness of angioplasty in moderate coronary stenosis: a randomized trial. Circulation. 2001 Jun 19;103(24):2928-34. doi: 10.1161/01.cir.103.24.2928. PMID 11413082
- [Background] Ahmadi A, Argulian E, Leipsic J, Newby DE, Narula J. From Subclinical Atherosclerosis to Plaque Progression and Acute Coronary Events: JACC State-of-the-Art Review. J Am Coll Cardiol. 2019 Sep 24;74(12):1608-1617. doi: 10.1016/j.jacc.2019.08.012. PMID 31537271
- [Background] McClelland RL, Jorgensen NW, Budoff M, Blaha MJ, Post WS, Kronmal RA, Bild DE, Shea S, Liu K, Watson KE, Folsom AR, Khera A, Ayers C, Mahabadi AA, Lehmann N, Jockel KH, Moebus S, Carr JJ, Erbel R, Burke GL. 10-Year Coronary Heart Disease Risk Prediction Using Coronary Artery Calcium and Traditional Risk Factors: Derivation in the MESA (Multi-Ethnic Study of Atherosclerosis) With Validation in the HNR (Heinz Nixdorf Recall) Study and the DHS (Dallas Heart Study). J Am Coll Cardiol. 2015 Oct 13;66(15):1643-53. doi: 10.1016/j.jacc.2015.08.035. PMID 26449133
- [Background] Fernandez-Friera L, Penalvo JL, Fernandez-Ortiz A, Ibanez B, Lopez-Melgar B, Laclaustra M, Oliva B, Mocoroa A, Mendiguren J, Martinez de Vega V, Garcia L, Molina J, Sanchez-Gonzalez J, Guzman G, Alonso-Farto JC, Guallar E, Civeira F, Sillesen H, Pocock S, Ordovas JM, Sanz G, Jimenez-Borreguero LJ, Fuster V. Prevalence, Vascular Distribution, and Multiterritorial Extent of Subclinical Atherosclerosis in a Middle-Aged Cohort: The PESA (Progression of Early Subclinical Atherosclerosis) Study. Circulation. 2015 Jun 16;131(24):2104-13. doi: 10.1161/CIRCULATIONAHA.114.014310. Epub 2015 Apr 16. PMID 25882487
- [Background] Ostgren CJ, Soderberg S, Festin K, Angeras O, Bergstrom G, Blomberg A, Brandberg J, Cederlund K, Eliasson M, Engstrom G, Erlinge D, Fagman E, Hagstrom E, Lind L, Mannila M, Nilsson U, Oldgren J, Ostenfeld E, Persson A, Persson J, Persson M, Rosengren A, Sundstrom J, Swahn E, Engvall JE, Jernberg T. Systematic Coronary Risk Evaluation estimated risk and prevalent subclinical atherosclerosis in coronary and carotid arteries: A population-based cohort analysis from the Swedish Cardiopulmonary Bioimage Study. Eur J Prev Cardiol. 2021 Apr 23;28(3):250-259. doi: 10.1177/2047487320909300. Epub 2020 Mar 3. PMID 33891684
- [Background] Gorgulho B, Alves MA, Teixeira JA, Santos RO, de Matos SA, Bittencourt MS, Bensenor I, Lotufo P, Marchioni DM. Dietary patterns associated with subclinical atherosclerosis: a cross-sectional analysis of the Brazilian Longitudinal Study of Adult Health (ELSA-Brasil) study. Public Health Nutr. 2021 Oct;24(15):5006-5014. doi: 10.1017/S1368980020005340. Epub 2021 Jan 8. PMID 33413712
- [Background] Miname MH, Bittencourt MS, Moraes SR, Alves RIM, Silva PRS, Jannes CE, Pereira AC, Krieger JE, Nasir K, Santos RD. Coronary Artery Calcium and Cardiovascular Events in Patients With Familial Hypercholesterolemia Receiving Standard Lipid-Lowering Therapy. JACC Cardiovasc Imaging. 2019 Sep;12(9):1797-1804. doi: 10.1016/j.jcmg.2018.09.019. Epub 2018 Nov 15. PMID 30448145
- [Background] Pagidipati NJ, Peterson ED. Should Cardiovascular Preventive Therapy Be Over-the-Counter? J Am Coll Cardiol. 2021 Sep 14;78(11):1124-1126. doi: 10.1016/j.jacc.2021.07.020. No abstract available. PMID 34503681